CLINICAL TRIAL: NCT02047812
Title: The Hospital Volume Relationship in Emergency Laparotomy Outcomes
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Other Study IDs: XRB13069-VEL
Record Dates: First submitted 2013-12-16; First posted 2014-01-28 (Estimated); Last update posted 2024-05-21 (Actual); Status verified 2014-01

CONDITIONS: Abdomen, Acute
Keywords: Laparotomy; General Surgery; Hospitals,General; Hospitals,High-Volume; Hospitals,Low-Volume; Outcome Assessment (Health Care)
MeSH Terms: conditions — Abdomen, Acute

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Biospecimen Retention: None Retained — Please note with regard to enrollment: that although this study period has ended and data is being collated, the actual number of subjects is not known at this point since data has yet to be received. We requested data on all subjects meeting our criteria within the time frame mentioned.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- High volume hospitals: The hospitals in the upper tertile for procedural volume
- Medium volume hospitals: The hospitals in the middle tertile for procedural volume
- Low volume hospitals: The hospitals in the lowest tertile for procedural volume.

SUMMARY:
Introduction

'Emergency Laparotomy' is an umbrella term for a set of commonly performed procedures which are known to carry a significant risk of mortality and morbidity. Previous work has shown considerable inter-hospital variation in emergency laparotomy outcomes within the United Kingdom. It is unknown whether there are significant differences in outcomes following laparotomy which may be explained by differences in hospital procedural volume.

Aims

The aim of this study is to compare emergency laparotomy outcomes in Scotland as they vary by hospital procedural volume.

Methods

This research study is a retrospective observational enquiry which will utilise administrative data from the Information Services Division (ISD) of NHS National Services Scotland. Patient episodes will be identified by a set of procedure codes for emergency laparotomy.

The primary outcome measure will be risk-adjusted 30 day/inpatient mortality, and secondary outcome measures will be 30 day readmission rate, 30 day re-operation rate and length of stay.

DETAILED DESCRIPTION:
The aim of this study is to explore the possibility of a hospital procedural volume-outcome relationship in Scottish emergency laparotomy outcomes.

This is a retrospective study of all emergency laparotomies performed in Scotland during the period from 1st January 2001 - 31st December 2010. It will use routinely collected administrative data from the Information Services Division (ISD) of NHS National Services Scotland.

Emergency laparotomy will be defined as a non-elective abdominal procedure primarily on the gut tube; and such cases will be identified by the use of a set of procedural codes, which will be validated against local records.

The registry which will supply the data for this study is the Scottish Morbidity Record 01 (SMR01), the full title of which is the "General / Acute Inpatient and Day Case dataset" (see http://www.adls.ac.uk/nhs-scotland/general-acute-inpatient-day-case-smr01/?detail). SMR01 is collated and administered by ISD, and data submission is mandatory for all Scottish NHS providers of in-patient or day-case care. Approximately 1.4 million records are added each year. Diagnoses are coded according to International Classification of Diseases (ICD)-10 standards and procedures are coded according to the United Kingdom's Office of Population Census Statistics (OPCS) standards, the most current of which is version 4.5. The data quality in SMR01 is high and is assured by regular internal audits. In the 2010 audit of accuracy, Main Condition was recorded with an accuracy of 88% and Main Procedure was recorded with an accuracy of 94%.

Where data inconsistencies are identified in the extract supplied for this study, further clarification will be obtained where possible with ISD's data retrieval support team. Data completeness is very high in SMR01. However, where significant volumes of data are missing or unusable, the need for data imputation will be explored.

The study period was decided on pragmatically by a desire to provide an assessment of current practice, fully within the era of widely practised laparoscopic surgery.

A power calculation also suggested that this would provide an adequate sample size to demonstrate mortality differences. A recent paper showed 30 day mortality for emergency laparotomy to be 14.9% (Saunders DI, Murray D, Pichel AC, Varley S, Peden CJ. Variations in mortality after emergency laparotomy: the first report of the UK Emergency Laparotomy Network. Br J Anaesth. 2012 Sep 1;109(3):368-75.)

We decided that we wanted to be able to detect a mortality difference (absolute) of 2%. Alpha was specified as 0.05 and power 0.9. Using a chi-2 test in G Power 3.1.7, it was determined that a total N of 5221 was required to show this difference. In the study already cited, 35 hospitals submitted data on 3 months of practice, giving a total of 1853 patients. We extrapolated to estimate that one hospital completes 212 laparotomies per year. There are currently 31 adult surgical centres in Scotland, resulting in an estimate of 6,565 laparotomies per year. Even accepting the smaller size of Scottish hospitals, this demonstrates that a 10 year cohort should be more than adequate to detect a clinically significant difference in length of stay.

Hospitals will be placed into tertiles of high, medium and low volume, according to the number of procedures performed over the study period.

The study will compare risk-adjusted 30 day/in-patient mortality as the primary outcome, with secondary outcomes of 30 day re-admission rate, 30 day re-operation rate and post-operative length of stay. Potentially significant confounding variables such as age, gender, and co-morbidity will be studied for their predictive value in a univariate model and included in a multivariate model if they remain significant.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged 18 years or older who undergo emergency laparotomy within the study period

Exclusion Criteria:

* Patients who are non-resident in Scotland
* Multiple laparotomies on a single patient will not be counted as separate index events unless ≥6 months have passed between previous discharge and new hospital admission.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All Scottish adult residents undergoing emergency laparotomy during the study period
Sampling Method: Probability Sample
Enrollment: 40000 (Actual)
Dates: Start 2001-01; Primary Completion 2010-12 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Mortality | Either within 30 days of procedure, or during continuous in-patient stay (up to 12.5 years)
  Death as an in-patient or ≤30 days of procedure.
  This is a retrospective study using a complete national data set, with the first admission 12.5 years distant from the time of data collection, and the last admission 2.5 years prior to the time of data collection. The theoretical maximal length of stay is 12.5 years.
  Deaths will be recognised from SMR01 which is linked to the Registrar General's database of deaths.

SECONDARY OUTCOMES:
Post-operative length of stay | From date of laparotomy to date of discharge (whole days) - up to 12.5 years
  (Whole) days from date of laparotomy to date of discharge. B
  This is a retrospective study using a complete national data set, with the first admission 12.5 years distant from the time of data collection, and the last admission 2.5 years prior to the time of data collection. The theoretical maximal length of stay is 12.5 years.
Re-operation | Within the index admission (theoretically, up to a maximum of 12.5 years) or within 30 days of discharge
  The occurrence of an abdominal procedure either subsequent to laparotomy and within the index admission, or ≤30 days of discharge.
  As above, this is a retrospective study using a complete national data set, with the first admission 12.5 years distant from the time of data collection, and the last admission 2.5 years prior to the time of data collection. The theoretical maximal length of stay for the index admission is 12.5 years.
Re-admission | Within 30 days of index discharge
  Re-admission to any hospital specialty ≤30 days have elapsed since date of discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Ewen M Harrison, FRCS, PhD, Principal Investigator — University of Edinburgh
Locations (1):
- All Scottish NHS Hospitals, Multiple Locations, United Kingdom